CLINICAL TRIAL: NCT01155297
Title: Effect of Physical Training on Quality of Life, Functional Capacity, Pulse Wave Velocity and Biochemical Markers in Patients With Chronic Renal Failure on Conservative Treatment
Brief Title: Effect of PT on QL, FC, PWV and Biochemical Markers in CRF on Conservative Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: UPECLIN HC FM Botucatu Unesp (Other)
Responsible Party: Viviana Rugolo Oliveira e Silva, UPECLIN HC FM Botucatu Unesp
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: upeclin/HC/FMB-Unesp-45
Record Dates: First submitted 2010-06-29; First posted 2010-07-01 (Estimated); Last update posted 2010-07-01 (Estimated); Status verified 2010-06

CONDITIONS: Kidney Failure, Chronic; Resistance Training; Treatment
Keywords: Quality of Life; Biological Markers; Renal Insufficiency; Resistance Training; Exercise; Chronic Kidney Failure
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency; Motor Activity | interventions — Physical Conditioning, Human; Exercise; Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Group (Sham Comparator): At the control group, with 34 subjects, will be performed stretching and metabolic exercises. This group will make the assessments before and the reassessments after the end of the program.
  Interventions: Behavioral: Stretching and metabolic exercises
- Training group (Active Comparator): At the training group, with 34 subjects, will be performed stretching, physical training and resistance. This group will make the assessments before and the reassessments after the end of the program.
  Interventions: Behavioral: Physical training

INTERVENTIONS:
Behavioral: Physical training — The exercise program will be held three times a week and will have three stages: local and global stretching, aerobic exercise for 30 minutes ( with 50 and 60% of maximal heart rate) and strength training. The strength training will be done after assessment of one repetition maximum (1RM) and the prescription will be made with 50% load of 1RM, where the patient will hold three sets of 10-12 repetitions. Reassessments will be conducted monthly for readjustment of the charges. The duration of the training protocol will be six months.
  After completing this exercise program, patients will undergo a reassessment repeating the ET and reapplication of the SF-36, redone the collection of ADMA serum concentration.
  Other Names: Exercise Training; Intervention group
  Arms: Training group
Behavioral: Stretching and metabolic exercises — At the control group will be performed stretching and metabolic exercises and will make the assessments and the reassessments after the end of the program.
  Other Names: Pumping exercises; Control Group
  Arms: Control Group

SUMMARY:
Introduction: Chronic Kidney Disease (CKD) is considered an important public health problem, with prevalence of 9.6% in our population. The CKD has as main symptoms fatigue, muscle weakness and poor exercise tolerance, which directly contribute to physical inactivity and low mobility, increasing the risk of morbidity and mortality in CKD patients with significant impact on quality of life of these patients. Thus, patients with CKD have poor quality of life, high incidence of cardiovascular diseases, high prevalence of endothelial dysfunction, the consequent increase in arterial stiffness and serum concentration of asymmetric dimethylarginine (ADMA). It is believed that the conditioning of these patients may reduce cardiovascular risks and improve the quality of life. Aim of the study: Evaluate the impact of exercise training in relation to functional capacity, quality of life, pulse wave velocity and ADMA in patients with CKD on dialysis. Materials and methods: Is a randomized controlled study, with 34 CKD patients on conservative treatment, divided into control group (with stretching exercises and metabolic exercises) and training group, those undergoing physical training, aerobic and resistance during six months. Before and after exercise training, patients will be assessed using the SF-36 and IPAQ. Also be held assessment of pulse wave velocity, measurement of serum ADMA and spirometry testing. Statistical analysis consisted of t test for independent data or chi-square when appropriate.

DETAILED DESCRIPTION:
The CKD is currently regarded as an important worldwide public health problem. In the United States, approximately 10.8% of population has this disease (Sarnak et al 2003) and it is estimated that by 2015 about 40 million people in this country will develop chronic renal failure (BRONAS, 2009). In Brazil, epidemiological data are rare, but there is a study that there is a prevalence of 9.6% in the population (Bastos et al, 2009).

The skeletal muscles of patients with CKD may present structural alteration and degeneration of muscle fibers, contributing to reduction of strength and endurance. The use of steroid medications, malnutrition, hormonal and electrolyte abnormalities are also other elements (CHAN, CHEEMA, SINGH, 2007). These symptoms directly contribute to physical inactivity and low mobility, increasing the risk of morbidity and mortality in patients with CKD (MANSUR LIMA; NOVAES, 2007).

To measure the quality of life of CKD patient is needed to identify how and in which dimensions of this patient's life is being affected, for such investigation SF 36 is widely used (CATTAI et al, 2007). The SF-36 assesses quality of life for the individual analysis of physical, social, emotional and mental health. (Castro et al, 2003).

There are numerous ways to assess functional capacity, and the cardiopulmonary exercise test (ET), is a valuable method for. Involves the assessment of respiratory, metabolic and cardiovascular variables by measurement of pulmonary gas exchange during exercise and expression of functional assessment indices (SIERRA, 1997; Yasbek JR, 1998). The functional capacity or aerobic capacity is determined by obtaining the contents of maximal oxygen uptake (VO2 max) and ventilatory anaerobic threshold (BARROS NETO; Tebexreni; TAMBEIRO, 2001). Several studies bounce the importance of physical activity and indicate the benefits that this can bring to patients with CKD on dialysis. Smith and colleagues (2007) submitted their dialysis patients to an exercise protocol, consisting of heating, stretching and active and resistance exercises conducted in 24 sessions. They observed a significant improvement in blood pressure (BP) and heart rate (HR), as well as improved quality of life assessed using the SF-36.

Patients with CKD have a high prevalence of cardiovascular disease (CVD) including coronary dysfunction, peripheral vascular dysfunction and heart failure (CANZIANI, 2004). The CVD represent the leading cause of death for patients in early stages of CKD, with a rate of approximately 45% in patients that do not do dialysis (Abedin et al, 2010). Recent studies have shown that markers of arterial stiffness are important predictors of mortality and morbidity related to CVD in CKD patients (MOLLER et al, 2007). The arterial stiffening is a hallmark of the aging process, due to changes in wall structure of arteries and the consequent remodeling process that can be accelerated by metabolic disturbances arising from the CKD (Frimodt-MOLLER et al, 2008; PORAZKO et al, 2009 ).

The pulse wave velocity (PWV) is a valid instrument to assess arterial distensibility, is recognized as gold standard for measuring arterial stiffness, because it has good reproducibility, noninvasive and easy to perform (Di Iorio et al , 2009).

Mustata et al (2004) in their study evaluated arterial stiffness and insulin resistance in dialysis patients, aiming to measure the impact of aerobic training on these variables and obtained as response a significant decrease in the values of arterial stiffness after training.

Toussaint et al (2008) conducted a prospective study on the impact of cycling during dialysis in arterial stiffness patients with CKD and found a significant improvement after physical training compared with no exercise. With this study the authors speculated that the improvement in arterial compliance was related to enhanced NO bioavailability serum. The results of these studies are promising and suggest that exercise training can improve arterial compliance and reduces left ventricular hypertrophy in patients with CKD. Clearly, more research is needed in this area to confirm these findings in patients with CKD.

Abedin et al (2010) analyzing data from a controlled study, found a high prevalence of vascular calcification and arterial stiffness in pre-dialysis patients, showing a positive relationship between the progression of CKD and CVD.

The CKD and generalized vasculopathy, mentioned above are accompanied by endothelial dysfunction (COSTA-HONG et al, 2009). One of the causes of endothelial dysfunction is the inhibition of nitric oxide (NO), an important vasodilator and potent factor that opposes the atherogenesis. This inhibition occurs, among other causes, increased serum concentration of the substance asymmetric dimethylarginine (ADMA) that is present mainly in CVD and CKD (Mittermayer et al, 2005).

Oner - Iyidogan et al (2009) show a close relationship between increased values of ADMA and CKD, justified by the lack of excretion of this substance. In another study, Gibson et al (2008) analyzed patients with metabolic syndrome and found that they had low endogenous NO formation and high concentrations of circulating ADMA.

The patient with CKD generally along the disease develops insulin resistance, CHF and high concentration of ADMA (ONER-IYIDOGAN et al, 2009). However in our knowledge no study has evaluated the effect of physical exercise in the value of ADMA serum of this group.

The only work in our knowledge that evaluated the impact of physical training in patients at pre-dialysis, written by Boyce et al (1997), examined variables as renal function, blood pressure and cardiorespiratory endurance. They concluded that exercise training reduces blood pressure, increases aerobic capacity and muscle strength.

Moinuddin and Leehey (2008) reported that aerobic exercise and muscle training are a great benefit to CKD patients, improving the VO2max and muscle mass. Chan, & Singh Cheema (2007), after undergoing 12 weeks of high intensity exercise with progressive and resistance training during hemodialysis routine, obtained as a result increased muscle mass and strength and subsequent improvement in quality of life of these patients.

Given the importance of the topic and the fact that appropriate therapeutic slow the progression of dysfunction, reduce the suffering of patients and reduce costs to the national health system, sees the need to study the implementation of physical rehabilitation in patients with CKD who are not undergoing hemodialysis. Therefore, this study aims to evaluate the impact of exercise training in relation to functional capacity, quality of life, pulse wave velocity and ADMA in patients with CKD on conservative treatment.

This project is a randomized controlled study that will be developed at Clinic Hospital, at School of Medicine of Botucatu. The work is approved by the Ethics and Research committee and will be started after the informed and formal consent of patients.

The data collection will begin with an assessment of quality of life using the SF-36 validated in Brazil; application the short version of IPAQ Questionnaire to identify sedentary patients, evaluation the PWV and the functional capacity with a spirometry test (brand Cosmed K4b2, Rome, Italy).

This study will use the lab test that is already part of routine in our department for monitoring patients with CKD, as The Brazilian Guidelines for Chronic Kidney Disease recommend. Simultaneously will be collected a venous blood sample for measurement of serum ADMA.

The results will be recorded and submitted to statistical analysis. The baseline characteristics of the groups will be compared by t test for independent data or chi-square when appropriate. The behavior of the groups will be analyzed by t test for dependent samples.

ELIGIBILITY:
Inclusion Criteria: Patients over 18 years, diagnosed with Chronic Kidney Disease, stages II to IV, and that shows contraindications to exercise training

Exclusion Criteria: Patients unable to understand the procedures that will be performed, previous diagnosis of coronary artery disease, uncontrolled chronic hypertension (BP ≥ 150 x 100 mm Hg), ET positive for cardiac ischemia, patients with cancer, liver failure or chronic or acute infection.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 68 (Estimated)
Dates: Start 2010-06; Primary Completion 2011-05 (Estimated); Study Completion 2011-11 (Estimated)

PRIMARY OUTCOMES:
The impact of exercise training in relation to functional capacity, quality of life, pulse wave velocity and ADMA in patients with CKD on dialysis | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Viviana Silva, graduate, Principal Investigator — State University of São Paulo "Júlio de Mesquita Filho", Medicine School of Botucatu; Luis Cuadrado, Doctor, Study Director — State University of São Paulo "Júlio de Mesquita Filho", Medicine School of Botucatu
Locations (1):
- State University of São Paulo "Júlio de Mesquita Filho", Medicine School of Botucatu, Botucatu, São Paulo, Brazil